CLINICAL TRIAL: NCT02183402
Title: Relative Bioavailability of Digoxin After Co-administration of Multiple Oral Doses of Digoxin (0.25 mg qd) and Multiple Oral Doses of BI 1356 (5 mg qd) Compared to the Bioavailability of Multiple Oral Doses of Digoxin (0.25 mg qd) Alone in Healthy Male and Female Volunteers (an Open-label, Randomized, Two-way Crossover Clinical Phase I Study)
Brief Title: Pharmacokinetics, Safety and Tolerability of Digoxin With or Without Co-administration of BI 1356 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.29
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; Linagliptin

ARMS (2):
- Digoxin with BI 1356 (Experimental)
  Interventions: Drug: Digoxin; Drug: BI 1356
- Digoxin (Active Comparator)
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin
Drug: BI 1356
  Arms: Digoxin with BI 1356

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics, safety and tolerability of digoxin with and without co-administration of BI 1356. Additionally the steady state pharmacokinetics of BI 1356 when co-administered with digoxin will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females and males according to the following criteria: based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥ 18 and age ≤ 50 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g., HIV)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than five half-lives of the respective drug prior to administration or during the trial
* Use of drugs which could reasonably influence the results of the trial or that prolonged the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day) or inability to stop alcoholic beverages for 24 hours prior to dosing and up to the last sampling time point
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that was of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a corrected QT interval > 450 ms)
* A history of additional risk factors for torsade de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For female subjects:

* Pregnancy/positive pregnancy test, or planning to become pregnant during the study or within one month of study completion
* No adequate contraception during the study and until one month of study completion
* Lactation period

Exclusion criteria specific for this study:

* Bradycardia (< 50/min) or atrioventricular block (including I grade auriculoventricular (AV) block) at screening
* Creatinine clearance (Cockroft-Gault-Formula) < 80 mL/min at screening
* History of or actual thyroid dysfunction/disease, or basal thyroid-stimulating hormone (TSH) , free triiodothyronine (FT3), or free thyroxine (FT4) out of normal range at screening
* Any degree of hypokalemia, hypomagnesemia, or hypercalcemia at screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve in plasma at steady state over a uniform dosing interval τ) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
Cmax,ss (maximum measured concentration in plasma at steady state over a uniform dosing interval τ) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
CLR,ss (renal clearance at steady state) for digoxin | 0-2 h, 2-4 h, 4-8 h, 8-12 h, 12-24 h, 24-48 h, 48-72 h, 72-96 h, 96-120 h, and 120-144 h after drug last administration on day 11

SECONDARY OUTCOMES:
AUC0-∞,ss (area under the concentration-time curve of the analyte in plasma at steady state over the time interval from 0 extrapolated to infinity) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
AUC0-tz,ss (area under the concentration-time curve of the analyte in plasma at steady state over the time interval from 0 to the last quantifiable drug plasma concentration ) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
AUCt1-t2,ss (area under the concentration-time curve of the analyte in plasma at steady state over the time interval t1 to t2) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
tmax,ss (time from (last) dosing to the maximum measured concentration of the analyte in plasma at steady state) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
λz,ss (terminal rate constant of the analyte in plasma at steady state) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
t1/2,ss (terminal half-life of the analyte in plasma at steady state) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
MRTpo,ss (mean residence time of the analyte in the body after oral administration at steady state) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
CL/F,ss (apparent clearance of the analyte in plasma following extravascular administration at steady state) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
Cpre,ss (the pre-dose steady state concentration of the analyte immediately before administration of the next dose) for digoxin | pre-dose (-0:30) on days 1, 8, 9, 10, 11
Vz/F,ss (apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state) for digoxin | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
Aet1-t2,ss (amount of analyte that is eliminated in urine from the time point t1 to time point t2 under steady state conditions) for digoxin | 0-2 h, 2-4 h, 4-8 h, 8-12 h, 12-24 h, 24-48 h, 48-72 h, 72-96 h, 96-120 h, and 120-144 h after drug last administration on day 11
fet1-t2,ss (fraction of administered drug excreted unchanged in urine at steady state over the respective time interval, where t1 and t2 define beginning and end times of the time interval) for digoxin | 0-2 h, 2-4 h, 4-8 h, 8-12 h, 12-24 h, 24-48 h, 48-72 h, 72-96 h, 96-120 h, and 120-144 h after drug last administration on day 11
AUCτ,ss (area under the concentration-time curve in plasma at steady state over a uniform dosing interval τ) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
Cmax,ss (maximum measured concentration in plasma at steady state over a uniform dosing interval τ) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
tmax,ss (time from (last) dosing to the maximum measured concentration of the analyte in plasma at steady state) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
λz,ss (terminal rate constant of the analyte in plasma at steady state) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
t1/2,ss (terminal half-life of the analyte in plasma at steady state) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
MRTpo,ss (mean residence time of the analyte in the body after oral administration at steady state) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
CL/F,ss (apparent clearance of the analyte in plasma following extravascular ministration at steady state) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
Cpre,ss (the pre-dose steady state concentration of the analyte immediately before administration of the next dose) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
Vz/F,ss (apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state) for BI 1356 | before (-0:30) administration of digoxin, 0:30, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 24:00, 48:00, 72:00, 96:00, 120:00, and 144:00 hours after administration of digoxin
Incidence of Adverse Events | Up to 66 Days
Assessment of global tolerability by the investigator | Day 17 of each trial period